CLINICAL TRIAL: NCT01911455
Title: Double-Blind, Placebo-Controlled Proof of Concept Study in Youth With Fragile X Syndrome
Brief Title: Study of Acamprosate in Fragile x Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CIN001- Acamprosate in FX
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2020-03

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acamprosate (Active Comparator): The maximum dose of acamprosate to be used in this study is 666 mg three times daily (total 1998 mg/day) for subjects weight ≥ 50 kg and 1332mg for subjects that weigh < 50 kg.
  Interventions: Drug: acamprosate
- Placebo (Placebo Comparator): Placebo will be prescribed with the same frequency and duration as the acamprosate group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: acamprosate
  Other Names: Campral
  Arms: acamprosate
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this research study we want to understand the effectiveness of a drug treatment, acamprosate, for interfering symptoms (i.e., inattention/hyperactivity, social impairment) associated with Fragile X Syndrome (FXS).

DETAILED DESCRIPTION:
Each subject with FXS will receive 10 weeks of blinded treatment with acamprosate or matching placebo. After completion of the double-blind phase, all subjects will have an opportunity to receive acamprosate as part of the study procedures for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic confirmation of full mutation FXS
* Age ≥5 years and <23 years
* General good health as determined by physical exam, medical history and laboratory work up.

Exclusion Criteria:

* Use of more than two psychotropic medications (medications affecting behavior).
* Unstable dosing of any psychotropic medication (medication affecting behavior)
* Problems with kidney functioning
* Unstable seizure disorder
* Change in any anti-convulsant drug dosing in the 60 days prior to study entry
* Prior adequate treatment trial with acamprosate as determined by the study doctor
* Pregnant or lactating females

Ages: 5 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-Social Withdrawal subscale | Change from baseline to week 10
  The ABC is the gold standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials.

SECONDARY OUTCOMES:
Clinical Global Impressions- Improvement (CGI-I) | week 10
  The CGI-I global improvement item is a 7-point Likert scale designed to measure symptomatic change at a specific time as compared to baseline. CGI-I is a gold standard global measure of potential change with treatment in placebo-controlled pharmacotherapy trials in developmental disabilities.
Aberrant Behavior Checklist- Hyperactivity (ABC-H) | Change from baseline to week 10
  The ABC is the gold standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials.
Aberrant Behavior Checklist-Social Avoidance (ABC-SA) | Change from baseline to week 10
  The ABC is the gold standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Erickson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Elizabeth Berry-Kravis, MD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio